CLINICAL TRIAL: NCT01866930
Title: Phase 3 Open Label Study Evaluating the Efficacy and Safety of Pegylated Interferon Lambda-1a, in Combination With Ribavirin and Daclatasvir, for Treatment of Chronic HCV Infection With Treatment naïve Genotypes 1, 2, 3 or 4 in Subjects Co-infected With HIV
Brief Title: Efficacy and Safety Study of Pegylated Interferon Lambda-1a With Ribavirin and Daclatasvir, to Treat naïve Subjects With Chronic HCV Genotypes 1, 2, 3, and 4 Who Are Co-infected With HIV
Acronym: DIMENSION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision not based on any new unexpected safety findings or efficacy observations.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI452-032; 2012-003280-22 (EudraCT Number)
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-02

CONDITIONS: Chronic Hepatitis C Infection
MeSH Terms: interventions — peginterferon lambda-1a; daclatasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A: GT-2 or -3 HCV Treatment Naïve Subjects (Experimental): Pegylated Interferon Lambda 180 µg solution, injection subcutaneously once weekly for 24 weeks
  Ribasphere 200 mg tablets (800 mg per day: two 200 mg tablets in the morning and two 200 mg tablets in the evening) by mouth twice daily for 24 weeks
  Daclatasvir 30 mg, 60 mg, or 90 mg tablets (depending on concomitant HIV regimen) once daily for 12 weeks
  Interventions: Biological: Pegylated Interferon Lambda-1a; Drug: Daclatasvir (DCV); Drug: Ribasphere (RBV)
- Cohort B: GT-1 or -4 HCV Treatment Naïve Subjects (Experimental): Pegylated Interferon Lambda 180 µg solution, injection subcutaneously once weekly for 24 or 48 weeks
  Ribasphere 200 mg tablets, (1000 mg per day: two 200 mg tablets in the morning and three 200 mg tablets in the evening for subjects weighing <75 kg and 1200 mg per day: three 200 mg tablets in morning and three 200 mg tablets in evening for subjects weighing ≥75 kg) by mouth twice daily for 24 or 48 weeks
  Daclatasvir 30 mg, 60 mg, or 90 mg tablets (depending on concomitant HIV regimen) once daily for 12 weeks
  Interventions: Biological: Pegylated Interferon Lambda-1a; Drug: Daclatasvir (DCV); Drug: Ribasphere (RBV)

INTERVENTIONS:
Biological: Pegylated Interferon Lambda-1a
  Other Names: BMS-914143
Drug: Daclatasvir (DCV)
  Other Names: BMS-790052
Drug: Ribasphere (RBV)

SUMMARY:
To evaluate Sustained Virologic Response at post treatment Week 12 (SVR12)following treatment with Lambda/RBV/DCV in chronic HCV GT-1, -2, -3 or -4 subjects co-infected with HIV-1

DETAILED DESCRIPTION:
Study Classification: Safety/Efficacy and Pharmacokinetics/dynamics

GT=genotype

ELIGIBILITY:
Inclusion Criteria:

* HCV Genotype-1, -2, -3 or -4 treatment naïve;
* HCV RNA ≥10,000 IU/mL at screening;
* HIV-1 infection [(approximately 200 subjects receiving HAART, approximately 100 subjects not receiving highly active antiretroviral therapy (HAART)];
* For subjects receiving HAART, HIV RNA must be below <40 copies/mL at screening and <200 copies/mL for at least 8 weeks prior to screening;
* CD4 cell count at screening must be ≥100 cells/μL if receiving HAART or ≥350 cells/μL if not receiving HAART)
* Seronegative for Hepatitis B Surface Antigen (HBsAg)
* Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive. BMI=weight (kg)/[height (m)]2 at screening;
* Subjects with compensated cirrhosis are permitted, but the number of subjects will be capped at approximately 30%. If a subject does not have cirrhosis, a liver biopsy within 3 years prior to enrollment is required to demonstrate the absence of cirrhosis. If cirrhosis is present, any prior liver biopsy is sufficient. Fibroscan® or FibroTest are acceptable if performed within 1 year prior to treatment in countries where liver biopsy is not required prior to treatment and where non-invasive imaging tests are approved for staging of liver disease
* Subjects with mild to moderate hemophilia as defined as:

  1. Mild-factor level activity of 6-4% OR
  2. Moderate defined as factor level activity of 1-5%

Exclusion Criteria:

* Any evidence of liver disease other than chronic HCV;
* Subjects infected with human immunodeficiency virus (HIV-2);
* Diagnosed or suspected hepatocellular carcinoma;
* Decompensated liver disease;
* Presence of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within 12 weeks prior to study entry (AIDS-defining opportunistic infections as defined by the CDC, (CDC, JAMA 1993 Feb 10;269(6):729-30)
* Laboratory values: ANC <1.5 x 109 cells/L (<1.2 x 109 cells/L for Blacks), platelet count <90 x 109 cells/L, hemoglobin <11 g/dL for females, hemoglobin <12 g/dL for males;
* Subjects (receiving HAART) who had first initiated anti-retroviral therapy within last 8 weeks prior to Day 1; however, if changes are required to a subject's HAART regimen to meet the requirements of the protocol, these changes are allowed at the screening visit. Subjects should wait a minimum of 1 month prior to Day 1 after a repeat of HIV viral load has been confirmed, <40 copies/mL
* Subjects on Zidovudine (AZT), Didanosine (ddI), or Stavudine (d4T);
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Subjects with severe hemophilia (defined as <1% factor activity level)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (54):
- United States (13):
  - Inland Empire Liver Foundation, Rialto, California
  - University Of California San Francisco, San Francisco, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - University Of Colorado Denver & Hospital, Aurora, Colorado
  - University Of Colorado Denver, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Orlando Va Medical Center, Orlando, Florida
  - Emory Hospital Midtown Infectious Disease Clinic, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Mercy Medical Center, Baltimore, Maryland
  - Duke Clinical Research Institute, Durham, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Ut Southwestern Medical Center, Dallas, Texas
- Argentina (4):
  - Local Institution, Buenos Aires, Bs As, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Quilmes, Buenos Aires
  - Local Institution, Buenos Aires
- Belgium (2):
  - Local Institution, Antwerp
  - Local Institution, Brussels
- Canada (7):
  - University Of Alberta Hospitals, Edmonton, Alberta
  - St Pauls Hospital, Vancouver, British Columbia
  - Vancouver Id Reserach & Care Centre Society, Vancouver, British Columbia
  - Hamilton Health Sciences, Mcmaster Site, Hamilton, Ontario
  - Ottawa Hospital General Campus, Ottawa, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Mcgill University Health Centre (Muhc) Montreal Chest Institute, Montreal, Quebec
- France (4):
  - Local Institution, Le Kremlin-Bicêtre
  - Local Institution, Lyon
  - Local Institution, Paris
  - Local Institution, Pessac
- Germany (3):
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Hamburg
- Italy (5):
  - Local Institution, Antella (fi)
  - Local Institution, Brescia
  - Local Institution, Milan
  - Local Institution, Monza
  - Local Institution, Roma
- Mexico (4):
  - Local Institution, Ciudad Juárez, Chihuahua
  - Local Institution, León, Guanajuato
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
- Poland (2):
  - Local Institution, Lodz
  - Local Institution, Wroclaw
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Volgograd
- Spain (4):
  - Local Institution, Barcelona
  - Local Institution, Cartagena (Murcia)
  - Local Institution, Donosti-San Sebastian
  - Local Institution, Madrid
- United Kingdom (3):
  - Local Institution, London, Greater London
  - Local Institution, Brighton
  - Local Institution, London

REFERENCES:
- [Derived] Nelson M, Rubio R, Lazzarin A, Romanova S, Luetkemeyer A, Conway B, Molina JM, Xu D, Srinivasan S, Portsmouth S. Safety and Efficacy of Pegylated Interferon Lambda, Ribavirin, and Daclatasvir in HCV and HIV-Coinfected Patients. J Interferon Cytokine Res. 2017 Mar;37(3):103-111. doi: 10.1089/jir.2016.0082. Epub 2017 Feb 17. PMID 28282271
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 453 participants were enrolled in the study. 300 participants were randomized and received treatment. 153 participants were not randomized to a treatment group due to Adverse Event (3), withdrawal of consent (13), loss to follow-up (4), administrative reasons per sponsor (5), no longer met study criteria (105), or other reasons (23).
Groups:
- Cohort A: HCV GT-2 or GT-3: Participants with HCV (Genotype 2 or 3) and HIV co-infection were treated with Lambda/RBV/DCV for 12 weeks followed by Lambda/RBV for 12 weeks, for a total treatment duration of 24 weeks. Participants received 180μg of Lambda via subcutaneous injection, once weekly, 800 mg/day Ribavirin tablets, orally, twice daily, for a planned duration of 24 weeks. Participants were administered 30 mg Daclatasvir tablets, orally, once daily, for a maximum of 12 weeks. The total daily dose was 30, 60 or 90 mg depending on the HIV concomitant regimen. Participants were followed up for a duration of 24 weeks after 24 weeks of treatment.
- Cohort B: HCV GT-1 or GT-4: Participants with HCV (Genotype 1 or 4) and HIV co-infection were treated with Lambda/RBV/DCV for 12 weeks followed by Lambda/RBV for either 12 or 36 weeks. Participants were administered 180μg of Lambda via subcutaneous injection, once weekly, for a maximum of 48 weeks; body weight stratified dose of Ribavirin tablets, orally, twice daily, for maximum duration of 48 weeks (<75 kg, total dose was 1000 mg/day, weighing >=75 kg, total dose was 1200 mg/day); and 30 mg Daclatasvir tablets, orally, once daily, for a maximum of 12 weeks. The total daily dose was 30, 60 or 90 mg depending on the HIV concomitant regimen. Participants who achieved an extended rapid virologic response (eRVR) during initial 12 weeks were treated with Lambda/RBV for 12 weeks for total of 24 weeks. Participants who did not achieve eRVR during initial 12 weeks were treated with Lambda/RBV for 36 weeks for total of 48 weeks. Participants were followed up for a duration of 24 weeks after 24 or 48 weeks of treatment.
Period: Treatment Period
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Started | 104 | 196
Completed | 95 | 161
Not Completed | 9 | 35
Not completed — Other | 1 | 0
Not completed — Death | 0 | 2
Not completed — Poor/non compliance | 0 | 2
Not completed — No longer meets study criteria | 0 | 1
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Lack of Efficacy | 1 | 9
Not completed — Adverse Event | 4 | 12
Not completed — Lost to Follow-up | 1 | 1
Period: Follow-up Period
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Started | 102 (Includes 7 participants who re-joined from previous period to follow-up period) | 185 (Includes 24 participants who re-joined from previous period to follow-up period)
Completed | 96 | 176
Not Completed | 6 | 9
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 1 | 5
Not completed — No longer required per protocol | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4 | Total
Number analyzed (Participants) | 104 | 196 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (8.88) | 46.6 (7.76) | 45.6 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 40 | 68
  Male | 76 | 156 | 232
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 41 | 79 | 120
  Unknown or Not Reported | 53 | 106 | 159
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 18 | 24
  White | 93 | 171 | 264
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
HCV Genotype [Count of Participants; unit: Participants]
  HCV GT-1 | 0 | 149 | 149
  HCV GT-2 | 20 | 0 | 20
  HCV GT-3 | 83 | 0 | 83
  HCV GT-4 | 0 | 41 | 41
  Unknown | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response at Post-treatment Week 12 (SVR12)
Description: SVR12 was defined as HCV RNA less than lower limit of quantification (< LLOQ) (25 IU/mL; target detected or not detected) at follow-up week 12.
Time Frame: Follow-up week 12
Population: The analysis was performed in all treated subjects using modified intent-to-treat algorithm, where the numerator is based on subjects meeting the response criteria and the denominator is based on all treated subjects (Non-completer = Failure).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
Participants | 88 | 149

2. Secondary Outcome: Number of Participants With Rapid Virologic Response (RVR) and Extended Rapid Virologic Response (eRVR)
Description: RVR is defined as HCV RNA < LLOQ target not detected at Week 4 and eRVR defined as HCV RNA < LLOQ target not detected at Weeks 4 and 12
Time Frame: Treatment weeks 4 and 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
Participants
  RVR | 82 | 149
  eRVR | 80 | 138

3. Secondary Outcome: Number of Subjects With Sustained Virologic Response at Post-treatment Week 24 (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ (25 IU/mL; target detected or not detected) at 24 weeks post treatment.
Time Frame: Follow-up week 24
Population: The analysis was performed in all treated subjects using modified intent-to-treat algorithm (numerator is based on subjects meeting the response criteria and the denominator is based on all treated subjects (Non-completer = Failure). Data was not collected for any participants due to termination of the study.
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Treatment Emergent Cytopenic Abnormalities
Description: All treated participants were monitored for treatment emergent cytopenic abnormalities (anemia as defined by hemoglobin (Hb) < 10 g/dL, and/or neutropenia as defined by absolute neutrophil count (ANC) < 750 mm3 and/or thrombocytopenia as defined by platelets < 50,000/mm3) during the treatment period (Weeks 1, 2, 4, 6, 8, 12, 20, and 24, and at Weeks 28, 32, 36, 40, 44, and 48 for subjects requiring those visits).
Time Frame: After Day 1 to end of treatment; up to Weeks 24 or 48
Population: Analysis was performed in all treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
Participants | 4 | 15

5. Secondary Outcome: Number of Participants With On-treatment IFN-associated Flu-like or Musculoskeletal Symptoms
Description: All treated participants were monitored for IFN-associated Flu-like and Musculoskeletal symptoms. Flu-like symptoms were defined as pyrexia, chills, or pain. Musculoskeletal symptoms were defined as arthralgia, myalgia, or back pain. Subjects were monitored throughout the treatment period during the treatment period (After day 1 up to week 24, or After day 1 up to week 48 for subjects requiring those visits).
Time Frame: After Day 1 to end of treatment; up to Weeks 24 or 48
Population: Analysis was performed in all treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
Participants
  Musculoskeletal symptoms | 6 | 21
  Flu-like symptoms | 6 | 19

6. Secondary Outcome: Number of Participants Who Died or Experienced Severe Adverse Events (SAEs), Dose Reductions of Lambda or Discontinuation Due to Adverse Events (AEs)
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that. at any dose, results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: After Day 1 to end of treatment; up to Weeks 24 or 48
Population: The analysis included all treated subjects up to the end of the treatment period (Day 1 to week 24, or Day 1 to week 48 for subjects requiring those visits).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
Participants
  Deaths | 0 | 3
  SAEs | 6 | 12
  Lambda Dose Reduction | 4 | 19
  Discontinuation due to AEs | 4 | 13

7. Secondary Outcome: Number of Participants With Treatment-emergent Grade 3/4 Lab Abnormalities
Description: Grade 3/4 treatment-emergent lab abnormalities that occurred in >=5% of subjects in either cohort are reported. The analysis included all treated subjects up to the end of the treatment period (Day 1 to week 24, or Day 1 to week 48 for subjects requiring those visits). Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling. AST = Aspartate aminotransferase, ALT = Alanine aminotransferase.
Time Frame: After Day 1 to end of treatment; up to Weeks 24 or 48
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
Participants
  Total Bilirubin | 26 | 63
  AST | 10 | 13
  ALT | 2 | 10

8. Secondary Outcome: Mean Change in Absolute CD4 T Lymphocyte Count From Baseline to End of Treatment
Description: All treated participants were monitored for change in Absolute CD4 T Lymphocyte count from Baseline to the end of the treatment period. The mean change in each arm for all evaluable participants is reported in Cells/µL.
Time Frame: Day 1 to end of treatment; up to week 24 or week 48
Population: The analysis was performed in all evaluable treated participants.
Measure: Mean (95% Confidence Interval); unit: Cells/uL
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
Cells/uL | -42.4 [-85.86 to 1.09] | -104.9 [-128.74 to -81.04]

9. Secondary Outcome: Mean Percent Change in Absolute CD4 T Lymphocyte Count From Baseline to End of Treatment
Description: All treated participants were monitored for percent change in CD4 T Lymphocyte count from Baseline to the end of the treatment period. The mean percent change in each arm is presented for all evaluable participants.
Time Frame: Day 1 to end of treatment; up to week 24 or week 48
Population: The analysis was performed in all evaluable treated participants.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
Percent change | -4.0 [-10.32 to 2.24] | -13.4 [-18.91 to -7.98]

10. Secondary Outcome: Mean Change in Total Lymphocyte Count From Baseline to End of Treatment
Description: All treated participants were monitored for change in Total Lymphocyte Count from Baseline to the end of the treatment period. The mean change in each arm for all evaluable participants is reported in Cells/µL.
Time Frame: Day 1 to end of treatment; up to week 24 or week 48
Population: The analysis was performed in all evaluable treated participants.
Measure: Mean (95% Confidence Interval); unit: Cells/µL
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
Cells/µL | -0.38 [-0.50 to -0.25] | -0.50 [-0.56 to -0.43]

11. Secondary Outcome: Mean Percent Change in Total Lymphocyte Count From Baseline to End of Treatment
Description: All treated participants were monitored for percent change in Total Lymphocyte Count from Baseline to the end of the treatment period. The mean percent change in each arm is presented for all evaluable participants.
Time Frame: Day 1 to end of treatment; up to week 24 or week 48
Population: The analysis was performed in all evaluable treated participants.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
Percent change | -15.33 [-20.46 to -10.19] | -22.95 [-26.04 to -19.86]

12. Secondary Outcome: Mean Change in Platelet Count From Baseline to End of Treatment
Description: All treated participants were monitored for change in Platelet Count from Baseline to the end of the treatment period. The mean change in each arm for all evaluable participants (units of measurement = x10^9 cells/L).
Time Frame: Day 1 to end of treatment; up to week 24 or week 48
Population: The analysis was performed in all evaluable treated participants.
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
10^9 cells/L | 32.7 [24.62 to 40.84] | 33.3 [27.10 to 39.57]

13. Secondary Outcome: Mean Percent Change in Platelet Count From Baseline to End of Treatment
Description: All treated participants were monitored for percent change in Platelet Count from Baseline to the end of the treatment period. The mean percent change in each arm is presented for all evaluable participants.
Time Frame: Day 1 to end of treatment; up to week 24 or week 48
Population: The analysis was performed in all evaluable treated participants.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
Number analyzed (Participants) | 104 | 196
Percent change | 16.9 [12.53 to 21.20] | 20.1 [16.10 to 24.16]

ADVERSE EVENTS:
Time Frame: Day 1 to end of treatment; up to week 24 or week 48, SAE: within 30 days of discontinuation of dosing
Arm/Group | Cohort A: HCV GT-2 or GT-3 | Cohort B: HCV GT-1 or GT-4
All-Cause Mortality (participants affected / at risk) | 0/104 | 3/196
Serious Adverse Events (participants affected / at risk) | 6/104 | 12/196
Other Adverse Events (participants affected / at risk) | 70/104 | 159/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: HCV GT-2 or GT-3 (N=104) | Cohort B: HCV GT-1 or GT-4 (N=196)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Multi-Organ failure (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 2 (2)
Dysthymic disorde (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 2 (2) | 2 (2)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Secondary syphilis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: HCV GT-2 or GT-3 (N=104) | Cohort B: HCV GT-1 or GT-4 (N=196)
Aspartate aminotransferase increased (Investigations) | 8 (10) | 4 (16)
Weight decreased (Investigations) | 4 (5) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 10 (10)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 16 (16)
Headache (Nervous system disorders) | 10 (13) | 31 (39)
Injection site erythema (General disorders) | 0 (0) | 12 (12)
Asthenia (General disorders) | 22 (24) | 32 (34)
Influenza like illness (General disorders) | 8 (9) | 5 (6)
Fatigue (General disorders) | 9 (9) | 47 (53)
Pyrexia (General disorders) | 3 (4) | 13 (13)
Depressed mood (Psychiatric disorders) | 2 (2) | 14 (15)
Anxiety (Psychiatric disorders) | 4 (4) | 15 (15)
Depression (Psychiatric disorders) | 6 (7) | 18 (18)
Insomnia (Psychiatric disorders) | 16 (19) | 31 (31)
Irritability (Psychiatric disorders) | 15 (16) | 23 (24)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 30 (43)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 15 (15)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 12 (12)
Nausea (Gastrointestinal disorders) | 10 (11) | 36 (51)
Vomiting (Gastrointestinal disorders) | 4 (4) | 23 (32)
Jaundice (Hepatobiliary disorders) | 6 (6) | 10 (11)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (4) | 12 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (17) | 33 (35)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (10) | 27 (27)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 26 (28)
Decreased appetite (Metabolism and nutrition disorders) | 9 (10) | 24 (27)

LIMITATIONS AND CAVEATS:
The study was ended prematurely, giving few participants an opportunity to reach follow-up week 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.